CLINICAL TRIAL: NCT05961787
Title: LARGE-ONE: A Prospective, Multicenter, Randomized Controlled Trial of the Use of Drug-coating Balloons(DCB) or Drug-eluting Stents(DES) in the Treatment of Large Diameter Coronary Atherosclerotic Lesions
Brief Title: A Trial of DCB vs DES in the Treatment of de Novo Large Diameter Coronary Atherosclerotic Stenosis(LARGE ONE)
Acronym: LARGE-ONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-IC-ISR-026
Record Dates: First submitted 2022-12-06; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB ARM (Experimental): patients with large primary coronary artery lesions (3.0mm≤ vessel diameter ≤4.0mm, lesion length ≤35mm).
  Interventions: Device: SeQuent® Please drug coating balloon(DCB)，Firehawk family drug eluting stent(DES)
- DES ARM (Active Comparator): patients with large primary coronary artery lesions (3.0mm≤ vessel diameter ≤4.0mm, lesion length ≤35mm).
  Interventions: Device: SeQuent® Please drug coating balloon(DCB)，Firehawk family drug eluting stent(DES)

INTERVENTIONS:
Device: SeQuent® Please drug coating balloon(DCB)，Firehawk family drug eluting stent(DES) — Investigation on DCB vs DES on Symptomatic or silent ischemic coronary artery disease with indications for PCI
  * Lesions ≤35 mm in length (visual), diameter 3-4 mm.
  * A maximum of 2 target lesions on 2 major epicardial coronary target vessels can be treated during baseline procedure. (e.g., one target lesion on one target vessel, or two target lesions on the same target vessel but separated ≥ 15 mm; Or 1 target lesion on each of the target vessels)

SUMMARY:
For the treatment of primary large-diameter coronary atherosclerosis through percutaneous coronary intervention (PCI), the use of a drug balloon (DCB) is not inferior to the placement of a drug-eluting stent (Firehawk™ family).

* Large-diameter vessels were defined as vessels with a diameter of ≥3.00 mm and ≤ 4.0mm

ELIGIBILITY:
Inclusion Criteria:

CI1. Age of subject 18-75 years old;

CI2. The subject (or legal guardian) understands and provides written informed consent to the test requirements and treatment procedures prior to performing any specific tests or procedures in the study;

CI3. The subject is suitable for percutaneous coronary intervention (PCI);

CI4. The subject had symptomatic coronary artery disease with objective evidence or asymptomatic ischemia;

CI5. Subject is willing to submit to all subsequent evaluations required by the test protocol

Angiogragh Inclusion

AI1. At Maximum 2 target lesions with stenosis ≥50%, located in no more than 2 vessels with a visual reference vessel diameter (RVD) of ≥3.00 mm and ≤4.00 mm;

AI2. The length of the target lesion must be≤35 mm (visually) and can be covered by one study stent or drug balloon;

AI3. The first target lesion must be successfully predilated/pretreated without:

1. Vascular tears affecting hemodynamics (TIMI blood grade ≤2);
2. Coronary dissection classified as D, E and F(ARC);
3. Residual stenosis > 30% after lesion preparation;

Note: If Type C dissection occurs at lesion predilation/preparation, clinical investigators will determine whether the target lesion can be included based on the comprehensive situation of blood flow and patients risks . Type C dissection will be excluded from the OCT subgroup considering the risk of dissection extension for OCT operation.

AI4. The anatomical conditions of the coronary artery were appropriate, and the study instrument could be transported to the appropriate location of the target lesion.

Exclusion Criteria:

CE1. Subjects with clinical symptoms and/or ECG findings consistent with the diagnosis of acute ST-segment elevation myocardial infarction (STEMI) within 7 days;

CE2. Subject is known to be allergic to contrast agents (which cannot be fully pretreated) and/or concomitant medications required by the stent system or protocol (e.g., cobalt-chrome, platinum-chrome, stainless steel, rapamycin, paclitaxel and similar configuration compounds, drug coating carrier components, all P2Y12 receptor inhibitors, aspirin, etc.);

CE3. Planned surgical treatment within 6 months after baseline surgery;

CE4. Severe heart failure (NYHA Grade IV) or left ventricular ejection fraction <30% (ultrasound or left ventricular contrast);

CE5. Previous renal impairment: serum creatinine >2.0mg/dL; Or on dialysis;

CE6. Previous bleeding events (BARC III or V);

CE7. Subject is receiving or indication of long-term anticoagulant therapy ;

CE8. Subject has any of the following conditions (baseline assessment) :

* Other serious medical conditions that reduce subjects' life expectancy to less than 13 months (e.g., cancer, congestive heart failure);
* Subject has a current substance abuse problem (e.g., alcohol, cocaine, heroin, etc.);
* Subject plans to undergo surgical/intervention procedures that may result in non-compliance with protocol or confusing data interpretation;

CE9. Subject has a history of bleeding tendency, coagulation disorders or refusal of blood transfusion;

CE10. The subject is participating in a clinical trial of another investigational drug or device that does not meet its primary endpoint;

CE11. Subjects are scheduled to participate in another investigational drug or device clinical trial within 13 months of baseline procedure;

CE12. Subjects who intend to be pregnant within 13 months of baseline procedure (fertile and sexually active women should consent to use a reliable contraceptive method from screening to 13 months after baseline surgery);

CE13. Subjects are pregnant or breastfeeding (fertile women with pregnancy possibility should undergo a pregnancy test within 7 days prior to baseline surgery).

Angiogragh Exclusion

AE1. Plan to treat 3 or more target lesions;

AE2. Plan to treat more than 2 major epicardial vessels;

AE3. A single lesion to be treated cannot be covered by a single stent or a single drug balloon;

AE4. The subject had two target lesions in the same target vessel, and the distance between the two target lesions was ≤15mm (visual observation);

AE5. Target lesions were located in the left main trunk;

AE6. Target lesions were located within 3mm of the initial segment of the left anterior descending artery (LAD) or left circumflex artery (LCX).

AE7. Target lesions were located in a saphenous vein, artery or artificial bypass graft;

AE8. Target lesions need to be treated through a saphenous vein, artery or artificial bypass graft ;

AE9. Target lesion blood flow grade of TIMI 0/1 before guide wire passes through ;

AE10. Treatment of target lesions involves multi-stent strategy in complex lesions (e.g., bifurcated lesions require more than one stent);

AE11. Target lesions involve previously in-stent restenosis lesions or overlap with previously implanted stents;

AE12. Subject has unprotected left main coronary artery disease (>50% diameter stenosis);

AE13. Subjects have received PCI for any type of target lesion (e.g., balloon dilation, stent placement, balloon dissection, etc.) within 12 months before baseline;

AE14. Presence of thrombus or possible thrombus in the target lesion (visual);

AE15. The target lesions were moderate to severe calcification lesions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Value of Luminal loss at 13month post procedure | 13 months
  defined as the difference between the minimum lumen diameter in the lesion segment immediately after use of the study instrument and the minimum lumen diameter at 13 months angiographic follow up .

SECONDARY OUTCOMES:
Rate of Target Lesion Failure(TLF) | 30 days, 6 months, 1and 2 years
  defined as the composite of cardiac death, target vessel-related myocardial infarction (MI)*, or ischemia-driven target lesion revascularization (TLR)
Rate of Major Adverse Cardiac Events(MACE ) | 30 days, 6 months, 1and 2 years
  The composite of cardiac death, any MI or ischemia-driven TLR, and stent thrombosis myocardial infarction (MI)*, or ischemia-driven target lesion revascularization (TLR)
Value of Neointimal Volume: | 3 months post procedure
  the total volume bounded by the stent and the lumen within the segment of interest. It can be calculated using the formula: [= Stent Volume - Lumen Volume]
Value of Stent Volume | 3 months post procedure
  Based on Simpson's rule, the stent volume is calculated as the total volume bounded by the stent within the segment of interest. In the absence of neointimal hyperplasia, malapposition, and tissue protrusion, the stent volume corresponds to the lumen volume.
Value of Lumen Volume | 3 months post procedure
  Based on Simpson's rule, the total volume bounded by the lumen within the segment of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zheng, Doctoral, Study Director — Shanghai MicroPort Medical (Group) Co., Ltd.
Locations (1):
- Jining Medical University Affiliated Hospital, Jining, Shandong, China